CLINICAL TRIAL: NCT02724995
Title: Finding Genes for Rare Diseases
Status: Withdrawn | Type: Observational
Why Stopped: Responsible party left the university of kentucky without enrolling any participants
Sponsor: University of Kentucky (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0735-P1H
Record Dates: First submitted 2016-02-10; First posted 2016-03-31 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Rare Diseases
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will help the investigator understand the pathogenesis of different rare genetic conditions and to establish database of rare genetic databases. This would ultimately help to provide more accurate diagnosis through advanced genomic diagnostic testing and databases established from this study. This knowledge would in turn help in the clinical management of other affected family members and other individuals affected with similar conditions. Understanding of pathogenesis of the disease would also enable the investigator to develop targeted therapies for rare genetic diseases, and also to collaborate on the targeted therapy-related clinical trials.

The investigator plans to store the results of this study in databases. These results will be shared with other researchers or doctors, who research, diagnose or treat the individuals with similar diseases.

The investigator will only share the data that is collected and not the biological samples.

DETAILED DESCRIPTION:
This proposed study is designed identify for the genetic causes of rare diseases. This study does not involve the use of investigational medication or devices. No randomization will take place. Participants enrolled into the study will be asked to provide blood or saliva samples for DNA testing. Samples will be collected by one of two methods;

* If the participant has had a clinical genetic test performed, the results/data will be collected from the University of Kentucky (UK) clinical molecular pathology laboratory or from the medical records. If the cause of the disease is not identified on clinical genetic testing, the investigator will reanalyze the clinical genetic testing data or use the blood or saliva sample leftover from the clinical genetic testing for additional experiments using new methods to identify the cause of the disease.
* If no sample leftover from the clinical genetic testing is available, the investigator plans to collect about 2 teaspoons of blood or saliva from the participant at their first visit to the site.

This study plans to enroll 1000 participants from the University of Kentucky Medical Center.

The investigator plans to store any blood or saliva DNA samples collected for future research studies involving rare genetic diseases. The stored blood or saliva DNA samples will not be released to anyone outside the study.

Stored samples will be labeled with a unique study identifier and will be maintained in the investigator's research laboratory located at the University of Kentucky, Department of Pathology and Laboratory Medicine, 800 Rose Street, Lexington, KY 40536.

There is no limit on the length of time that the samples will be stored. The investigator may keep using the stored samples indefinitely unless the participant decide to withdraw from the project.

Participants may withdraw or cancel their permission for the use for their stored samples at any time. However, any samples and health information already obtained from their use will not be destroyed.

There will be no additional costs or charges to the participant for allowing the investigator to store and use their left over blood or saliva samples and there is no benefit to the participant for allowing the investigator to store their samples.

Participants will not be paid for donating their samples. The samples and information that the participants are donating will no longer belong to them. The research may lead to new medical knowledge, tests, treatments or products. These products could have some financial value. There are no plans to provide financial payment to either the participant or their relatives should this occur.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a rare genetic disease
* Are between the ages of 0 and 101
* Are willing to have genetic testing performed on blood or saliva samples
* Can understand and speak English

Exclusion Criteria:

* Diagnosis of cancer
* Unwilling to have genetic testing performed on blood or saliva samples
* Unable to read or speak English
* Prisoners

Ages: 1 Minute to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with rare genetic diseases
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Number of Rare Genetic Diseases Diagnosed using Advanced Genomic Technologies | 5 years
  Investigators will use genomic technologies such as SNP microarray, Array CGH, Whole exome and whole genome sequencing to identify the mutations causing different rare diseases. These results will be reported to the patients or parents after confirming in the CLIA certified laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Sivakumaran T Arumugam, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No